CLINICAL TRIAL: NCT00768326
Title: A Double-blind, Randomised, Parallel-group, Placebo-controlled Study of the Safety, Tolerability and Efficacy Following Sequential Dose Regimens of Lu 31-130 to Patients With Schizophrenia
Brief Title: Efficacy of Lu 31-130 in Patients With Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11613A; EudraCT 2006-003739-57 (Registry Identifier: EudraCT)
Record Dates: First submitted 2008-10-07; First posted 2008-10-08 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Antipsychotic; Lu 31-130
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Zicronapine. Study Part A (Experimental)
  Interventions: Drug: Zicronapine
- Zicronapine. Study Part B (Experimental)
  Interventions: Drug: Zicronapine
- Zicronapine. Study Part C (Experimental)
  Interventions: Drug: Zicronapine
- Zicronapine. Study Part D (Experimental)
  Interventions: Drug: Zicronapine
- Zicronapine. Study Part E (Experimental)
  Interventions: Drug: Zicronapine
- 2A, 2B, 2C, 2D, 2E (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zicronapine — Study Part A:
  3mg; orally, film-coated tablets, once daily, 8 weeks
  Other Names: Lu 31-130
  Arms: Zicronapine. Study Part A
Drug: Zicronapine — Study Part B:
  5mg; orally, film-coated tablets, once daily, 8 weeks
  Other Names: Lu 31-130
  Arms: Zicronapine. Study Part B
Drug: Zicronapine — Study Part C:
  7mg; orally, film-coated tablets, once daily, 8 weeks
  Other Names: Lu 31-130
  Arms: Zicronapine. Study Part C
Drug: Zicronapine — Study Part D:
  2 x 5mg; orally, film-coated tablets, once daily, 8 weeks
  Other Names: Lu 31-130
  Arms: Zicronapine. Study Part D
Drug: Zicronapine — Study Part E:
  2 x 7mg; orally, film-coated tablets, once daily, 8 weeks
  Other Names: Lu 31-130
  Arms: Zicronapine. Study Part E
Drug: Placebo — Study Part A, B, C, D and E:
  Placebo; orally, film-coated tablets, once daily, 8 weeks
  Arms: 2A, 2B, 2C, 2D, 2E

SUMMARY:
The main purpose with the study is to evaluate the efficacy and safety of Lu 31-130 in patients suffering from schizophrenia compared to placebo.

DETAILED DESCRIPTION:
Schizophrenia is a serious and disabling mental disorder that affects approximately 1% of the world's population. Antipsychotic drugs remain the cornerstone in the pharmacotherapy of schizophrenia. However, none of the available drugs is ideal, in particular because of their complex safety profile and the limited effectiveness against certain symptoms of the disease. Thus, only one dimension of the morbidity, that is, the positive symptoms, can be expected to respond to treatment whereas negative symptoms and cognitive deficits are, at best, only marginally targeted.

Given this, there is no doubt that the current antipsychotic drugs leave much room for improvement and call for new, more effective pharmacotherapies in the treatment of schizophrenia. In the current study, patients suffering from schizophrenia and experiencing clinically significant symptoms of the disease will be included. In the current study, eligible patients will be randomised in a 2:1 ratio to blinded treatment with either Lu 31-130 (3, 5, 7, 10 or 14 mg/day) or placebo for 8 weeks. The study includes 5 parts with increasing doses of Lu 31-130 (Part A [3 mg/day], B [5 mg/day], C [7 mg/day], D [10 mg/day], and E [14 mg/day]). A decision to initiate Part B [5 mg/day of Lu 31-130], C [7 mg/day of Lu 31-130] or D [10 mg/day of Lu 31-130] will be based on safety and tolerability of the previous study part. Dependent on the safety, tolerability and PK data from Part D the study may proceed with Part E. The efficacy and the safety of Lu 31-130 will be evaluated in comparison to the pooled placebo group from all 5 study parts.

ELIGIBILITY:
Inclusion Criteria:

* The patient has a primary diagnosis of schizophrenia
* The patient experiences clinically significant symptoms
* The patient did not experience an acute exacerbation requiring hospitalisation within the last 6 months
* The patient's medication has been stable for at least 4 weeks prior screening
* The subject has normal serum values of parameters associated with liver function

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2007-03; Primary Completion 2009-10 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Safety: Adverse events, clinical safety laboratory tests (including liver biochemistry tests), metabolic parameters (including blood lipids, blood glucose weight, waist circumference), abnormal movements | 8

SECONDARY OUTCOMES:
Efficacy: Change in the Positive and Negative Syndrome Scale (PANSS) score from baseline to Week 8 as compared to placebo, change from baseline in Clinical Global Impression/Improvement (CGI-S/I) scores as compared to placebo | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (1):
- DE001, Munich, Germany

REFERENCES:
- Available data/document: EMA EudraCT Results: 2006-003739-57 — https://www.clinicaltrialsregister.eu/ctr-search/trial/2006-003739-57/results